CLINICAL TRIAL: NCT00316589
Title: A Multicenter, Open-label, Controlled Phase II Study to Evaluate Safety and Immunogenicity of MVA-BN® (IMVAMUNE) Smallpox Vaccine in 18-55 Year Old Naive and Previously Vaccinated HIV Infected Subjects With CD4 Counts >200 - 750/µl.
Brief Title: Safety and Immunogenicity of IMVAMUNE® (MVA-BN®) Smallpox Vaccine in HIV Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POX-MVA-011
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: HIV Infections
Keywords: HIV; treatment experienced; treatment vaccinia naive
MeSH Terms: conditions — HIV Infections | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy subjects (Experimental): Control group with and without a history of previous smallpox vaccination IMVAMUNE (MVA-BN)
  Interventions: Biological: IMVAMUNE (MVA-BN)
- HIV-infected, vaccinia-naive (Experimental): Subjects without a history of previous smallpox vaccination, IMVAMUNE (MVA-BN)
  Interventions: Biological: IMVAMUNE (MVA-BN)
- HIV-infected, vaccinia-experienced (Experimental): Subjects with a history of previous smallpox vaccination, IMVAMUNE (MVA-BN)
  Interventions: Biological: IMVAMUNE (MVA-BN)

INTERVENTIONS:
Biological: IMVAMUNE (MVA-BN) — 2 immunizations, four weeks apart: 1 x 10E8 TCID50, subcutaneous
  Other Names: IMVANEX

SUMMARY:
The purpose of this study is to gather information on the safety and immunogenicity of an investigational smallpox vaccine in HIV infected populations. Subjects will receive two vaccinations

ELIGIBILITY:
* Genders eligible for Study: Both
* Age: between 18 and 55 years
* Healthy volunteers are accepted

Inclusion Criteria:

* Subjects tested positive for HIV-1 infection (HIV-infected subjects).
* Subjects that are tested negative for HIV (Healthy subjects).
* Either on stable antiretroviral therapy or not on antiretroviral therapy.
* CD4 cells > = 200 - 750/µl.
* Subjects must be in good general health except for HIV infection.
* Women must not be pregnant and use an acceptable method of contraception.

Exclusion Criteria:

* Impairment of immunologic function (other than HIV infection).
* History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure.
* Uncontrolled serious infection.
* History of or active autoimmune disease.
* History or clinical manifestation of clinically significant and severe hematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders.
* History of an immediate family member (father, mother, brother, or sister) who has had onset of ischemic heart disease before the age of 50 years.
* High risk of developing a myocardial infarction or coronary death.
* History of intravenous drug abuse (within the last 12 months).
* Known allergy to egg or aminoglycoside (gentamicin).
* History of anaphylaxis or severe allergic reaction.
* Subjects undergoing treatment for tuberculosis infection or disease.
* Chronic administration of systemic immuno-suppressants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 581 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Turner Overton, MD, Principal Investigator — Washington University School of Medicine
Locations (36):
- United States (34):
  - Alabama Vaccine Research Clinic; University of Alabama at Birmingham, Birmingham, Alabama
  - Health for Life Clinic, PLLC, Little Rock, Arkansas
  - Providence Clinical Research, Burbank, California
  - Northern California Research, Carmichael, California
  - CSI Clinical Trials, Inc., Fountain Valley, California
  - AltaMed Health Services, Los Angeles, California
  - Alta Bates Summit Medical Center, East Bay AIDS Center, Oakland, California
  - Benchmark Clinical Research, San Francisco, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Consultive Medicine, Daytona Beach, Florida
  - Northpoint Medical, PA, Fort Lauderdale, Florida
  - The Kinder Medical Group, Miami, Florida
  - Infectious Diseases of NW Florida, Pensacola, Florida
  - Palm Beach Center, West Palm Beach, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - The CORE Center, Chicago, Illinois
  - Northstar Medical Center, Chicago, Illinois
  - Indiana University School of Medicine; Division of Infectious Disease, Indianapolis, Indiana
  - University of Iowa, Division of Infectious Diseases, Iowa City, Iowa
  - Nemechek Health Renewal, Kansas City, Missouri
  - St. Louis University, Center for Vaccine Dev., St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Immuniodeficiency Clinic, ECMC, Buffalo, New York
  - Universtity of Rochester School of Medicine, Rochester, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, Pittsburgh, Pennsylvania
  - Brown Medical School, Providence, Rhode Island
  - University of South Carolina, Columbia, South Carolina
  - Vanderbilt University, AIDS Clinical Trials Center, Nashville, Tennessee
  - Nicholaos C. Bellos, MD PA, Dallas, Texas
  - Valley AIDS Council, Harlingen, Texas
  - Diversified Medical Practices, Houston, Texas
- Puerto Rico (2):
  - Clinical Research P.R., Inc., San Juan
  - Maternal Infant Studies Center (CEMI), San Juan

REFERENCES:
- [Result] Overton ET, Stapleton J, Frank I, Hassler S, Goepfert PA, Barker D, Wagner E, von Krempelhuber A, Virgin G, Meyer TP, Muller J, Badeker N, Grunert R, Young P, Rosch S, Maclennan J, Arndtz-Wiedemann N, Chaplin P. Safety and Immunogenicity of Modified Vaccinia Ankara-Bavarian Nordic Smallpox Vaccine in Vaccinia-Naive and Experienced Human Immunodeficiency Virus-Infected Individuals: An Open-Label, Controlled Clinical Phase II Trial. Open Forum Infect Dis. 2015 May 5;2(2):ofv040. doi: 10.1093/ofid/ofv040. eCollection 2015 Apr. PMID 26380340

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy naïve: Healthy, smallpox vaccine-naïve subjects
- HIV naïve: HIV-infected, smallpox vaccine-naïve subjects
- Healthy Experienced: Healthy, smallpox vaccine-experienced subjects
- HIV Experienced: HIV-infected, smallpox vaccine-experienced subjects
Period: Overall Study
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Started (Vaccinated) | 88 | 352 | 9 | 132
Completed (active study period) | 87 | 328 | 8 | 127
Not Completed | 1 | 24 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 1
Not completed — Subject unwilling/unable to comply | 0 | 6 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Other reason | 0 | 12 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced | Total
Number analyzed (Participants) | 88 | 351 | 9 | 131 | 579
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (7.14) | 36.8 (7.98) | 45.6 (8.88) | 44.6 (5.13) | 37.5 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 64 | 4 | 21 | 139
  Male | 38 | 287 | 5 | 110 | 440
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 0 | 27 | 0 | 7 | 34
  United States | 88 | 324 | 9 | 124 | 545

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Incidence, relationship and intensity of any Serious Adverse Event (SAE)
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 88 | 351 | 9 | 131
Participants
  Any SAE | 0 | 17 | 0 | 6
  Any SAE with intensity >= Grade 3 | 0 | 15 | 0 | 5
  Any SAE assessed as related to vaccine | 0 | 1 | 0 | 0

2. Secondary Outcome: Related Grade >=3 Adverse Events
Description: Incidence of any Grade 3 or higher adverse drug reaction (missing, unknown, not evaluable, possibly, probably, or definitely related) to the study vaccine
Time Frame: within 29 days after any vaccination
Population: Full Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 88 | 351 | 9 | 131
Participants | 7 | 26 | 0 | 5

3. Secondary Outcome: Solicited Local Adverse Events
Description: Incidence and intensity of solicited local AEs (pain, erythema, swelling). Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 88 | 351 | 9 | 131
Participants
  Pain: Any | 79 | 246 | 7 | 79
  Pain: Grade >=3 | 9 | 28 | 1 | 4
  Erythema: Any | 68 | 160 | 7 | 61
  Erythema: Grade >=3 | 2 | 1 | 0 | 0
  Swelling: Any | 56 | 139 | 6 | 52
  Swelling: Grade >=3 | 1 | 1 | 0 | 0

4. Secondary Outcome: Solicited General Adverse Events
Description: Incidence of solicited general AEs (increased body temperature, headache, myalgia, chills, nausea, and fatigue): Intensity and relationship to vaccination. Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 88 | 351 | 9 | 131
Participants
  Increased body temperature: Any | 9 | 26 | 1 | 15
  Increased body temperature: Related | 5 | 17 | 1 | 11
  Increased body temperature: Grade >=3 | 0 | 2 | 0 | 0
  Headache: Any | 40 | 117 | 1 | 29
  Headache: Related | 29 | 86 | 0 | 17
  Headache: Grade >=3 | 5 | 11 | 0 | 5
  Myalgia: Any | 30 | 122 | 1 | 35
  Myalgia: Related | 28 | 100 | 1 | 26
  Myalgia: Grade >=3 | 4 | 11 | 0 | 3
  Chills: Any | 12 | 58 | 0 | 11
  Chills: Related | 6 | 42 | 0 | 7
  Chills: Grade >=3 | 0 | 3 | 0 | 1
  Nausea: Any | 15 | 52 | 0 | 22
  Nausea: Related | 12 | 42 | 0 | 12
  Nausea: Grade >=3 | 3 | 7 | 0 | 4
  Fatigue: Any | 28 | 108 | 2 | 40
  Fatigue: Related | 22 | 84 | 1 | 29
  Fatigue: Grade >=3 | 2 | 11 | 0 | 3

5. Secondary Outcome: Unsolicited Adverse Events: Incidence
Description: Incidence of any unsolicited adverse events
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 88 | 351 | 9 | 131
Participants | 59 | 236 | 3 | 73

6. Secondary Outcome: Unsolicited Adverse Events: Intensity
Description: Occurrence of unsolicited adverse events by Intensity
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Number; unit: events
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 88 | 351 | 9 | 131
events
  Total | 149 | 590 | 6 | 175
  Grade 1 | 113 | 410 | 3 | 134
  Grade 2 | 32 | 143 | 2 | 28
  Grade 3 | 4 | 34 | 1 | 13
  Grade 4 | 0 | 3 | 0 | 0
  Missing | 0 | 0 | 0 | 0

7. Secondary Outcome: Unsolicited Adverse Events: Relationship to Vaccination
Description: Occurrence of unsolicited adverse events by relationship to study vaccine
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Number; unit: events
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 88 | 351 | 9 | 131
events
  Unrelated/None | 45 | 236 | 0 | 87
  Unlikely | 40 | 167 | 1 | 42
  Possible | 22 | 109 | 1 | 23
  Probable | 16 | 45 | 1 | 12
  Definite | 26 | 31 | 3 | 11
  Missing | 0 | 2 | 0 | 0
  Total | 149 | 590 | 6 | 175

8. Secondary Outcome: CD4+ T-cell Counts
Description: Median CD4+ T-cell counts over time
Time Frame: within 32 weeks
Population: Full Analysis Set (HIV infected subjects)
Measure: Median (Full Range); unit: CD4 count (cells/µL)
Arm/Group | HIV naïve | HIV Experienced
Number analyzed (Participants) | 351 | 131
CD4 count (cells/µL)
  Week 0 | 445.0 [156 to 1108] | 456.0 [186 to 922]
  Week 1 | 434.5 [147 to 2029] | 455.0 [136 to 1107]
  Week 6 | 438.5 [125 to 1045] | 447.0 [213 to 1081]
  Week 32 | 403.5 [138 to 1056] | 435.0 [273 to 762]

9. Secondary Outcome: CD8+ T-cell Counts
Description: Median CD8+ T-cell counts over time
Time Frame: within 32 weeks
Population: Full Analysis Set (HIV infected subjects)
Measure: Median (Full Range); unit: CD8 count (cells/µL)
Arm/Group | HIV naïve | HIV Experienced
Number analyzed (Participants) | 351 | 131
CD8 count (cells/µL)
  Week 0 | 771.0 [62 to 3210] | 877.5 [188 to 1914]
  Week 1 | 779.0 [208 to 3449] | 848.0 [219 to 2066]
  Week 6 | 749.0 [177 to 3238] | 798.5 [229 to 2319]
  Week 32 | 834.0 [196 to 2457] | 729.0 [245 to 1870]

10. Secondary Outcome: Viral Load
Description: Viral load (HIV-1 RNA levels) over time
Time Frame: within 32 weeks
Population: Full Analysis Set (HIV infected subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | HIV naïve | HIV Experienced
Number analyzed (Participants) | 351 | 131
Participants
  Week 0: Missing | 13 | 5
  Week 0: <400 | 262 | 112
  Week 0: 400 - <1000 | 11 | 3
  Week 0: 1000 - <10000 | 42 | 6
  Week 0: >=10000 | 23 | 5
  Week 1: Missing | 15 | 7
  Week 1: <400 | 257 | 113
  Week 1: 400 - <1000 | 13 | 2
  Week 1: 1000 - <10000 | 44 | 5
  Week 1: >=10000 | 22 | 4
  Week 6: Missing | 31 | 10
  Week 6: <400 | 240 | 105
  Week 6: 400 - <1000 | 18 | 3
  Week 6: 1000 - <10000 | 41 | 6
  Week 6: >=10000 | 21 | 7
  Week 32: Missing | 275 | 108
  Week 32: <400 | 59 | 22
  Week 32: 400 - <1000 | 5 | 0
  Week 32: 1000 - <10000 | 4 | 1
  Week 32: >=10000 | 8 | 0

11. Secondary Outcome: PRNT Seroconversion Rate
Description: Seroconversion rate based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (6) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Per-protocol set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 57 | 241 | 5 | 91
percentage of subjects
  Week 1 | 5.3 [1.1 to 14.6] | 14.5 [10.3 to 19.6] | 60.0 [14.7 to 94.7] | 45.1 [34.6 to 55.8]
  Week 4 | 17.5 [8.7 to 29.9] | 21.6 [16.6 to 27.3] | 60.0 [14.7 to 94.7] | 62.6 [51.9 to 72.6]
  Week 6 | 78.9 [66.1 to 88.6] | 58.1 [51.6 to 64.4] | 80.0 [28.4 to 99.5] | 76.9 [66.9 to 85.1]
  Week 8 | 78.9 [66.1 to 88.6] | 52.7 [46.2 to 59.1] | 80.0 [28.4 to 99.5] | 78.0 [68.1 to 86.0]
  Week 32 | 16.7 [5.6 to 34.7] | 12.5 [5.2 to 24.1] | 60.0 [14.7 to 94.7] | 64.7 [38.3 to 85.8]

12. Secondary Outcome: PRNT GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Titers below the detection limit are included with a value of '1'.
Time Frame: within 32 weeks
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 57 | 241 | 5 | 91
Titer
  Week 0 | 1.3 [1.0 to 1.8] | 2.0 [1.6 to 2.4] | 12.0 [0.7 to 205.6] | 5.5 [3.6 to 8.4]
  Week 1 | 1.6 [1.1 to 2.4] | 2.9 [2.2 to 3.7] | 108.9 [2.9 to 4150.0] | 20.5 [12.6 to 33.4]
  Week 4 | 2.1 [1.3 to 3.3] | 3.7 [2.8 to 4.9] | 100.2 [2.7 to 3721.7] | 42.3 [26.9 to 66.4]
  Week 6 | 20.8 [12.3 to 35.3] | 13.0 [9.6 to 17.5] | 354.5 [66.2 to 1899.2] | 88.9 [59.2 to 133.5]
  Week 8 | 14.8 [9.2 to 24.0] | 9.7 [7.2 to 12.9] | 171.2 [62.2 to 470.9] | 76.1 [52.0 to 111.4]
  Week 32 | 2.8 [1.2 to 6.3] | 3.3 [2.0 to 5.6] | 58.0 [11.1 to 303.2] | 53.1 [27.2 to 103.7]

13. Secondary Outcome: ELISA Seroconversion Rate
Description: Seroconversion rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Per-protocol set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 57 | 241 | 5 | 91
percentage of subjects
  Week 1 | 24.6 [14.1 to 37.8] | 29.5 [23.8 to 35.7] | 80.0 [28.4 to 99.5] | 58.2 [47.4 to 68.5]
  Week 4 | 80.7 [68.1 to 90.0] | 69.3 [63.1 to 75.1] | 100.0 [47.8 to 100.0] | 79.1 [69.3 to 86.9]
  Week 6 | 98.2 [90.6 to 100.0] | 97.1 [94.1 to 98.8] | 100.0 [47.8 to 100.0] | 94.5 [87.6 to 98.2]
  Week 8 | 96.5 [87.9 to 99.6] | 92.1 [88.0 to 95.2] | 100.0 [47.8 to 100.0] | 90.1 [82.1 to 95.4]
  Week 32 | 66.7 [47.2 to 82.7] | 46.4 [33.0 to 60.3] | 60.0 [14.7 to 94.7] | 76.5 [50.1 to 93.2]

14. Secondary Outcome: ELISA GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Titers below the detection limit are included with a value of '1'.
Time Frame: within 32 weeks
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 57 | 241 | 5 | 91
Titer
  Week 0 | 1.9 [1.2 to 3.0] | 4.6 [3.5 to 6.0] | 37.1 [2.6 to 529.8] | 33.3 [21.5 to 51.5]
  Week 1 | 3.7 [2.1 to 6.5] | 9.4 [6.9 to 12.8] | 260.6 [36.6 to 1858.0] | 89.9 [56.0 to 144.3]
  Week 4 | 56.2 [34.9 to 90.5] | 46.6 [35.7 to 60.9] | 461.1 [63.8 to 3332.9] | 220.1 [154.5 to 313.5]
  Week 6 | 526.2 [400.2 to 691.8] | 299.8 [253.4 to 354.7] | 612.9 [107.6 to 3490.5] | 588.4 [463.6 to 746.7]
  Week 8 | 312.9 [235.5 to 415.8] | 175.5 [143.6 to 214.6] | 403.4 [77.0 to 2112.0] | 453.1 [370.7 to 553.7]
  Week 32 | 32.1 [14.7 to 70.1] | 24.3 [12.7 to 46.5] | 89.5 [3.6 to 2230.7] | 203.9 [152.7 to 272.4]

15. Secondary Outcome: ELISPOT IFN-γ: Response Rate
Description: Response rate based on number of subjects with response in an interferon gamma (IFN-γ) ELISPOT assay. Response is defined as the appearance of a signal in subjects that had no signal at Baseline or a relative increase by a factor of ≥1.7 compared to Baseline in subjects that had a signal at Baseline. Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Elispot Analysis Set (subset of the Per-protocol Set with ELISPOT data available)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 23 | 35 | 3 | 68
percentage of subjects
  Week 1 | 39.1 [19.7 to 61.5] | 28.6 [14.6 to 46.3] | 0.0 [0.0 to 70.8] | 26.5 [16.5 to 38.6]
  Week 4 | 39.1 [19.7 to 61.5] | 20.0 [8.4 to 36.9] | 33.3 [0.8 to 90.6] | 29.4 [19.0 to 41.7]
  Week 6 | 47.8 [26.8 to 69.4] | 40.0 [23.9 to 57.9] | 0.0 [0.0 to 70.8] | 29.4 [19.0 to 41.7]
  Week 8 | 30.4 [13.2 to 52.9] | 25.7 [12.5 to 43.3] | 0.0 [0.0 to 70.8] | 29.4 [19.0 to 41.7]
  Week 32 | 52.4 [29.8 to 74.3] | 36.8 [16.3 to 61.6] | 50.0 [1.3 to 98.7] | 23.1 [5.0 to 53.8]

16. Secondary Outcome: ELISPOT IFN-γ: SFU
Description: Median number of interferon gamma (IFN-γ) secreting peripheral blood mononuclear cells (PBMC) in response to stimulation with MVA-BN detected by ELISPOT assay.
Time Frame: within 32 weeks
Population: Elispot Analysis Set (subset of the Per-protocol Set with ELISPOT data available)
Measure: Median (Full Range); unit: Spot Forming Units / 10^6 PBMC
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
Number analyzed (Participants) | 23 | 35 | 3 | 68
Spot Forming Units / 10^6 PBMC
  Week 0 | 0.0 [0 to 230] | 0.0 [0 to 239] | 155.0 [88 to 542] | 0.0 [0 to 233]
  Week 1 | 87.0 [0 to 497] | 0.0 [0 to 806] | 71.0 [0 to 322] | 0.0 [0 to 375]
  Week 4 | 93.0 [0 to 501] | 0.0 [0 to 371] | 569.0 [100 to 1143] | 0.0 [0 to 603]
  Week 6 | 99.0 [0 to 754] | 72.0 [0 to 822] | 54.0 [0 to 751] | 57.5 [0 to 570]
  Week 8 | 0.0 [0 to 599] | 0.0 [0 to 505] | 71.0 [0 to 96] | 53.0 [0 to 550]
  Week 32 | 71.0 [0 to 942] | 73.0 [0 to 370] | 596.0 [454 to 738] | 0.0 [0 to 365]

ADVERSE EVENTS:
Arm/Group | Healthy naïve | HIV naïve | Healthy Experienced | HIV Experienced
All-Cause Mortality (participants affected / at risk) | 0/88 | 1/351 | 0/9 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/88 | 17/351 | 0/9 | 6/131
Other Adverse Events (participants affected / at risk) | 51/88 | 172/351 | 3/9 | 45/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy naïve (N=88) | HIV naïve (N=351) | Healthy Experienced (N=9) | HIV Experienced (N=131)
Neurosyphilis (Infections and infestations) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchitis acute (Infections and infestations) | 0 | 1 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anticonvulsant toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy naïve (N=88) | HIV naïve (N=351) | Healthy Experienced (N=9) | HIV Experienced (N=131)
Diarrhoea (Gastrointestinal disorders) | 2 | 14 | 0 | 6
Nausea (Gastrointestinal disorders) | 2 | 9 | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Injection site bruising (General disorders) | 2 | 2 | 0 | 0
Injection site nodule (General disorders) | 3 | 6 | 1 | 0
Injection site pain (General disorders) | 2 | 3 | 0 | 0
Injection site pruritis (General disorders) | 22 | 66 | 2 | 22
Injection site warmth (General disorders) | 2 | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 8 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 10 | 0 | 1
Sinusitis (Infections and infestations) | 5 | 6 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 7 | 0 | 2
Electrocardiogram abnormal (Investigations) | 2 | 2 | 0 | 0
Troponin I increased (Investigations) | 9 | 31 | 0 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 12 | 0 | 2
Headache (Nervous system disorders) | 5 | 8 | 0 | 3
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 12 | 1 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 4
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes